CLINICAL TRIAL: NCT05938374
Title: Preoperative Moderately Fractionated Intensity-modulated Radiotherapy (IMRT) With/Without Concurrent Fluzoparil for Locally Extremity or Trunk Sarcoma
Brief Title: Preoperative Moderately Fractionated IMRT for Locally Extremity or Trunk Sarcoma (SPARE-03)
Acronym: SPARE-03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, NINGNING LU, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC-4016
Record Dates: First submitted 2023-06-21; First posted 2023-07-10 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Soft Tissue Sarcoma
Keywords: soft tissue sarcoma; preoperative radiotherapy; moderately fractionated RT; Complications; PARP inhibitor
MeSH Terms: conditions — Sarcoma | interventions — fluzoparib

STUDY DESIGN:
Intervention Model Description: Preoperative moderately fractionated RT with Fluzoparib Preoperative moderately fractionated RT without Fluzoparib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative moderately fractionated RT with Fluzoparib (Experimental): Patients will receive preoperative moderately fractionated radiotherapy (RT)(43.5Gy/15fr). One week before RT onset, during radiotherapy and 5 weeks post-RT, patients also take oral Fluzoparib (100mg, BID, five days per week).
  Wide resection surgery would be done around 6 -10 weeks post-RT.
  Interventions: Drug: Fluzoparib; Radiation: Preoperative moderately fractionated radiotherapay
- Preoperative moderately fractionated RT without Fluzoparib (Experimental): Patients will receive preoperative moderately fractionated radiotherapy (RT)(43.5Gy/15fr). No radio-sensitizing drugs was given.
  Wide resection surgery would be done around 6 -10 weeks post-RT.
  Interventions: Radiation: Preoperative moderately fractionated radiotherapay

INTERVENTIONS:
Drug: Fluzoparib — One week before RT onset, during radiotherapy and 5 weeks post-RT, patients also take oral Fluzoparib (100mg, BID, five days per week).
  Other Names: RT+Fluzoparib
  Arms: Preoperative moderately fractionated RT with Fluzoparib
Radiation: Preoperative moderately fractionated radiotherapay — Patients will receive preoperative moderately fractionated radiotherapy (RT)(43.5Gy/15fr).
  Other Names: RT

SUMMARY:
To investigate the safety and efficacy of preoperative moderately fractionated IMRT and concurrent Fluzoparib Hydrochloride for primary truncal or extremity soft tissue sarcoma.

DETAILED DESCRIPTION:
To investigate the safety and efficacy of preoperative moderately fractionated IMRT and concurrent Fluzoparib Hydrochloride for primary truncal or extremity soft tissue sarcoma; To investigate the Quality of life and extremity function post-combination treatment; To study the mechanism of radio-sensitizing effects of Fluzoparib Hydrochloride for primary truncal or extremity soft tissue sarcoma; To assess the relationship between the MRI imaging, pathological findings and local control.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years.
* Histology proven soft tissue sarcoma of truncal or extremity, deemed appropriate for preoperative radiotherapy and conservative surgery by multidisciplinary discussion.
* ECOG 0-3
* Histology reviewed by reference pathologist
* Lesion can be assessed
* Can tolerate radiotherapy and Fluzoparib (Fluzoparib group)
* Agree contraception.
* Informed consent: All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed

Exclusion Criteria:

* No gross tumor post-resection in other center.
* Contraindications to Fluzoparib, including allergic to Fluzoparib, active bleeding, ulcer, enteric perforation, enteric obstruction, uncontrolled hypertension, Grade 3 to 4 cardiac insufficiency (per NYHA criteria), and severe hepatic or renal insufficiency (Grade 4), etc.
* Dermatofibrosarcoma protuberans(DFSP), Desmoids, etc.
* Benign histology
* Secondary cancer within 5 years (except cervical carcinoma in situ or early-stage skin basal cell carcinoma)
* STS can be cured by extensive operation alone.
* Previous irradiation to the same area
* radiological evidence of distant metastases
* Other contraindications, can't tolerate operation or other treatment needed in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Major wound complications | 4-months post-surgery
  Number of Participants with Major wound complications 4 months post-surgery

SECONDARY OUTCOMES:
Acute toxicities | pre-IMRT, weekly during IMRT, at the end of IMRT, 1 months post-IMRT
  acute toxicities were evaluated as per CTCAE V5.0 criteria weekly during IMRT and 1 months after IMRT
Late toxicities | 6 months, 9 months, 12 months, 18 months and 24 months after surgery
  late toxicities were evaluted as per CTCAE V5.0 criteria and RTOG scale after 6 months
Quality of Life | pre-IMRT, end of IMRT, 1 months post-IMRT, and then 3 months, 6 months, 9 months, 12 months, 18 months and 24 months after surgery
  EORTC QLQ-C30 questionnaire
Extremity function | pre-IMRT, end of IMRT, 1 months post-IMRT, and then 3 months, 6 months, 9 months, 12 months, 18 months and 24 months after surgery
  MSTS questionnaire, TESS questionnaire
Pathological complete remission rate | 2 weeks after surgery
  No residual tumor cells were observed on post-operative specimens
2-year overall survival | 2 year since enrollment
  Incidence of participants who were alive
2-year local control | 2 year since enrollment
  Incidence of participants who had no Local relapse

CONTACTS AND LOCATIONS:
Overall Officials: Ning-Ning Lu, Dr., Principal Investigator — Cancer Hospital and Institute, National Cancer Center, CAMS& PUMC, Beijing, China
Locations (2):
- China (2):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Cancer Hospital and Institute, National Cancer Center, Chinese Academy of Medical Sciences & Peking Union Medical Center, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided